CLINICAL TRIAL: NCT05158400
Title: Diagnostic Value of Hand Ultrasound in Assessment of Rheumatoid Arthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Fady Boles Anwer, resident doctor at Diagnostic and Interventional Radiology, Sohag university, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med-21-12-04
Record Dates: First submitted 2021-12-12; First posted 2021-12-15 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Patient's With Rheumatoid Arthritis
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cases (Experimental)
  Interventions: Radiation: Ultrasound

INTERVENTIONS:
Radiation: Ultrasound — Ultrasound examination on the hand

SUMMARY:
Rheumatoid arthritis (RA) is one of the most common autoimmune rheumatic diseases, affecting one in 100 individuals worldwide. It is considered a complex systemic multifactorial inflammatory process in which the immune system targets synovial joints and causes mild to severe joint destruction with extra-articular manifestations.

If left untreated, RA leads to deformity, considerable disability, and major comorbid conditions, including cardiovascular disease and increased mortality.

Early treatment with targeted therapies can alter long-term outcomes by minimizing disease activity, preventing joint damage and disability, and improving patients' quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Adult-onset disease.
2. Patients who fulfill the 2010 American College of Rheumatology/European League Against Rheumatism classification criteria for rheumatoid arthritis.

Exclusion Criteria:

1. Any patient with any collagen disease rather than Rheumatoid arthritis.
2. Patients with joints deformities.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-12-15 (Estimated); Primary Completion 2022-03-15 (Estimated); Study Completion 2022-03-15 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of Ultrasound in Rheumatoid Arthritis of the hand | 3 months
  detecting hand ultrasound findings in 30 patients with clinical manifestations suggesting Rheumatoid Arthritis (including synovial thickening, joint effusion, tenosynovitis, bone erosions) particularly in early disease activity, reporting the collected data to assess aspects of strength and weakness of ultrasound use in those patients

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaeley GS, Bakewell C, Deodhar A. The importance of ultrasound in identifying and differentiating patients with early inflammatory arthritis: a narrative review. Arthritis Res Ther. 2020 Jan 2;22(1):1. doi: 10.1186/s13075-019-2050-4. PMID 31898524
- [Background] Tan YK, Ostergaard M, Conaghan PG. Imaging tools in rheumatoid arthritis: ultrasound vs magnetic resonance imaging. Rheumatology (Oxford). 2012 Dec;51 Suppl 7:vii36-42. doi: 10.1093/rheumatology/kes329. PMID 23230093
- [Background] Rowbotham EL, Grainger AJ. Rheumatoid arthritis: ultrasound versus MRI. AJR Am J Roentgenol. 2011 Sep;197(3):541-6. doi: 10.2214/ajr.11.6798. PMID 21862794